# Official title of the study: Emotional state among patients with neurological disorders

### **Primary Investigator:**

Evgenia Trevlaki

Academic Fellow of International Hellenic University

NCT number: Not available

**Date**: 07/04/2022

## **Study protocol**

| Title | Emotional state among patients with neurological disorders |
|---|---|
| Methodology | cross-sectional observational study |
| Study Duration | through study completion, an average of 1 year |
| Study Center(s) | |
| Number of | Approximately 100 subjects |
| Subjects | |
| Diagnosis and | <ul> <li>Adults (&lt;18 years) with neurological deficit</li> </ul> |
| Main Inclusion | Admitted less than a week |
| Criteria | Able to speak |
| 0. 1.5.1. | |
| Study Product, | |
| Dose, Route, | |
| Regimen | |
| Statistical | Statistical analysis was conducted using the SPSS software (CI 95%) for |
| Methodology | descriptive statistics of the sample and for Statistical Significance evaluation. |
| | More specifically, Mann Whitney U and Kruskal Wallis tests were used to explore the relationships developed between the demographic and clinical |
| | characteristics with the DASS-21 variables scoring, while at the same time |
| | chi-square tests were performed to obtain a better understand of the |
| | sample's identity. |

#### **Background/introduction:**

#### Purpose:

This study tries to identify how demographic and clinical characteristics affect the patients DASS-21 scoring.

#### Methods:

Study Design.

This study is a cross-sectional observational study, which allow us to calculate the frequency of depression, anxiety, and stress in patients with Neurologic disorders and whether it is a risk factor for the progression of the disease.

Study population and selection criteria

The research took place in a private physiotherapy practice and 12 patients form the sample.

Data collection and reporting

Statistical analysis was conducted using the SPSS software (CI 95%) for descriptive statistics of the sample and for Statistical Significance evaluation. More specifically, Mann Whitney U and Kruskal Wallis tests were used to explore the relationships developed between the demographic and clinical characteristics with the DASS-21 variables scoring, while at the same time chi-square tests were performed to obtain a better understand of the sample's identity.

| Results |
|------------|
| Discussion |
| Conclusion |
| References |